CLINICAL TRIAL: NCT03315585
Title: The Efficacy and Safety of Composite Steep-pulse Treatment Apparatus Used in Prostate Cancer Focal therapy-a Phase I Study
Brief Title: The Efficacy and Safety of Composite Steep-pulse Treatment Apparatus Used in Prostate Cancer Focal Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Second Military Medical University (Other)
Responsible Party: Principal Investigator, yinghao Sun, director, head of uroglogy department, clinical professor, Second Military Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REMD-FA2017001
Record Dates: First submitted 2017-07-02; First posted 2017-10-20 (Actual); Last update posted 2018-04-13 (Actual); Status verified 2018-04

CONDITIONS: Prostate Cancer
Keywords: focal therapy; IRE; Composite Steep-pulse Treatment Apparatus; prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Steep Pulse Device (Experimental): Applying the steep pulse to treat the patients with Prostate cancer
  Interventions: Device: steep pulse device

INTERVENTIONS:
Device: steep pulse device — Applying the steep pulse to treat the patients with Prostate cancer

SUMMARY:
This trial is studying the effects and safety in treating patients with local prostate cancer with a new IRE device called Composite Steep-pulse Treatment Apparatus. This new device could cause cell irreversible electroporation, which leading necrosis of tumor cells. It also has the ability to prevent nerve,vessel, urethral and capsule unnecessary injury beside the ablation area. Composite Steep-pulse Treatment Apparatus will be used in patients who pass inclusion/exclusion criteria. Safety, quality of life, and histopathological analysis of prostate speciem will be evaluated in each study patients.

DETAILED DESCRIPTION:
Background:

Prostate cancer is the most common cancer in elderly males in western country. It is also a major health concern, especially in China with its greater proportion of elderly men in the general population. Currently, radical prostatectomy(RP) is the mainstream treatment for localized PCa to show a benefit for cancer-specific survival (CSS). However, the patient who underwent RP might suffer from the complication of erectile dysfunction or urinary incontinence. In 2004, a new method using steep pulses to treat tumor was appeared. It showed that steep pulses could bring about Irreversible Electroporation (IRE) of cell, leading tonecrosis of tumor cells. And it seemed to do no harms to the nerve and Vascular epithelial cell. The device of steep pulse had already been approved by FDA in 2011.However, this device of steep pulse has disadvantages like: (1)sever muscle contraction;(2)Urethral injury; (3)Capsule injury;(4)Nerve degeneration. This new device which is called Composite Steep-pulse Treatment Apparatus, may have the potential to conquer these disadvantages.

Purpose:

1. This study will assess the efficacy of Composite Steep-pulse Treatment Apparatus in the treatment of PCa.
2. This study will assess potency, urinary continence and complication rate for the patients undergo the treatment with steep pulse device.
3. Histopathological analysis of prostate speciem 4 weeks after treated by Composite Steep-pulse Treatment Apparatus.

Methods:

1. patients recruitment
2. transperineal prostate targeted biopsy guided by multiparametric magnetic resonance imaging/transrectal ultrasound (mpMRI/TRUS) fusion, plus systemic prostate biopsy.
3. Frozen pathological analysis will be performed;
4. Irreversible Electroporation of malignant Tumor Cell under Composite Steep-pulse Treatment for the patients with positive biopsy;
5. Complication, urinary continence, and sexual function will be evaluated after the IRE treatment;
6. RP for these patients in 4 weeks after the treatment of Composite Steep-pulse Treatment.
7. Histopathological Outcomes analysis will be performed to evaluate tumor residual rate, urethral injuries, nerve injuries and capsule injury in and beside the ablation area.

ELIGIBILITY:
Inclusion Criteria:

1. Prostate MRI can identify the suspect region(pi-RADS≥4 ) ,and no evidence of lymphatic metastasis
2. Patients must have confirmed prostate cancer by prostate biopsy
3. There must be no evidence of metastatic disease as confirmed by ECT and whole-body MRI
4. No prostatic calculus or prostatic calculus≤5mm
5. No contraindication on total intravenous anesthesia
6. Not take any anticoagulants before or discontinue anticoagulant therapy at least 7 days
7. Age ≥ 30 - ≤ 75 years
8. Life expectancy of greater than 10 years
9. Patients scheduled for radical prostatectomy.
10. Sexually potent

Exclusion Criteria:

1. Patients have previously undergone radical prostatectomy.
2. Patients have previously undergone hormonal therapy or radiotherapy.
3. Patients underwent other surgery before less than 3 months
4. Clinically significant cardiovascular disease
5. Patients with other malignant tumor or patients with hiv.
6. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
7. Patients with poor health condition
8. Simultaneous participation in another clinical trial

Ages: 30 Years to 75 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-04-27 (Actual); Primary Completion 2017-10-27 (Actual); Study Completion 2017-10-27 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] of IRE(with Composite Steep-pulse Treatment Apparatus) ablation procedure | 1 Year
  To determine if the IRE(with Composite Steep-pulse Treatment Apparatus) ablation procedure is safe as measured by the composite number of procedural, device and post procedural adverse events measured with the CTCAE proforma.
Efficacy (persentage of unablated tissue un the ablation zone) | 1 month
  Persentage of normal glandular tissue in the specified targeted ablation zone by histopathology assessment

SECONDARY OUTCOMES:
Sexual function | 1 month
  Mean sexual function domain score (IIEF-5 scoring:
  The IIEF-5 score is the sum of the ordinal responses to the 5 items. 22-25: No erectile dysfunction 17-21: Mild erectile dysfunction 12-16: Mild to moderate erectile dysfunction 8-11: Moderate erectile dysfunction 5-7: Severe erectile dysfunction)
Urinary incontinence | 1 month
  Mean urinary incontinence domain score (the number of pad everyday,good is less than 2 pads a day, more or equal than 2 pads a day)

CONTACTS AND LOCATIONS:
Overall Officials: yinghao sun, MD,PHD, Principal Investigator — Changhai Hospital
Locations (1):
- Changhai Hospital,Second Military Medical University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided